CLINICAL TRIAL: NCT06133868
Title: The Efficacy of Lavender and Chamomile Essential Oils Inhalation in Management of Dental Anxiety and Pain in Children Undergoing Local Anesthesia Administration and Primary Tooth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: clinical professor (Unknown)
Responsible Party: Principal Investigator, Sara Ibrahim Mansour Elsherbini, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Lavander vs chamomile
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anxiety, Dental
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental group) Chamomile (Active Comparator): - · Describing the method for the child to become familiar with
  · The patient will inhale natural chamomile oil in a separate room prior to the intervention. Three drops (0.1 cc per drop) will be poured on a cotton roll, and patients will inhale the oil without skin contact for 3 min.
  Interventions: Drug: Lavender and Chamomile Essential Oils
- - Group II (Experimental group) Lavender (Active Comparator): * Describing the method for the child to become familiar with.
  * The patient will inhale natural lavender oil (100% pure Lavandula) in a separate room prior to the intervention. Three drops (0.1 cc per drop) of lavender oil will be poured on a cotton roll, and patients will inhale the oil without skin contact for 3 min
  Interventions: Drug: Lavender and Chamomile Essential Oils
- - Group III (Control group) Cotton with saline (Placebo Comparator): * Describing the method for the child to become familiar with
  * The patient will inhale a clear cotton roll with saline.
  Interventions: Drug: Lavender and Chamomile Essential Oils

INTERVENTIONS:
Drug: Lavender and Chamomile Essential Oils — essential oils

SUMMARY:
The Efficacy of Lavender and Chamomile Essential Oils Inhalation in Management of Dental Anxiety in Children Undergoing Local Anesthesia Administration and Primary Tooth Extraction.

DETAILED DESCRIPTION:
Dental anxiety refers to an atypical and excessive fear of seeking dental care for preventative purposes or treatment, as well as an unreasonable level of anxiety in relation to dental operations. According to reports, dental anxiety frequently leads to elevated levels of caries and behavioral management difficulties in children. Furthermore, it has been observed that they exhibit impaired oral function and compromised oral esthetics. In the context of pediatric dentistry, several stimuli such as visual cues (e.g., needles), auditory cues (e.g., drilling sounds), olfactory cues (e.g., scents of cut dentin and eugenol), and tactile cues (e.g., high frequency vibrations) commonly contribute to the provoking of anxiety .

Aromatherapy is a form of complementary medicine where the use of essential oils has been found to contribute to the improvement of emotional well-being, the promotion of tranquillity, and the induction of relaxation in the human body . Aromatherapy has attracted interest in the dentistry area because to its alternative nature, since it is considered a possible method for preventative and analgesic purposes. This entails the application of vital aromatic compounds through the methods of inhalation, massage, or ingestion.

Lavender oil is widely recognized as a prominent fragrant oil within the field of aromatherapy, renowned for its anxiolytic properties The calming qualities of lavender oil have been historically acknowledged, making it a highly effective essential oil in the realm of aromatherapy. According to an article titled "Effect of Lavender Oil on Anxiety" it has been shown that lavender oil possesses stimulating properties on the parasympathetic system, leading to a subsequent decrease in both blood pressure and levels of anxiety. Multiple investigations have elucidated the existence of pharmacological actions with sedative properties, which exhibit dose-dependent characteristics. Furthermore, the incorporation of supplements exhibiting these benefits has recently been introduced into clinical practice .

Moreover, Kreidel et al., in 2021, suggested that lavender oil can be safely inhaled as a kind of aromatherapy, as no adverse effects have been reported. Therefore, the administration of lavender oil through inhalation is widely regarded as the most secure method among all available options. In their study. , it was determined that aromatherapy has the potential to serve as a non-aversive approach, wherein patients are exposed to pleasant aromas during dental procedures. Due to the favorable outcomes observed in medical contexts and among adult dental patients, a considerable number of dental professionals hold the belief that employing these methodologies could be efficacious in the treatment of children dental patients.

. Abd Alkhalek et al. (2023) examined the effects of lavender and orange essential oil inhalation on children's vital signs and anxiety during dental treatment. The study comprised 60 children who needed primary tooth extractions. Lavender, Orange, and Control oils were inhaled by the children. Before treatment, the patient's pulse, blood pressure, and oxygen saturation were checked. After the essential oil inhalation, anaesthetic, and extraction, measurements were taken. The Wong Baker Scale measured child anxiety. The Lavender and Orange groups showed a statistically significant reduction in anxiety levels after therapy, according to the Wong Packer Pain Scale. Heart rate and breathing rate also decreased. The experiments showed lavender outperformed orange.

Chamomile is a further medicinal plant employed in the practice of aromatherapy . Chamomile essential oil, derived from the herbaceous plant belonging to the Asteraceae family, is one of the several oils that can be effectively used in the practice of inhalation aromatherapy. Apigenin, a chemical included in chamomile, demonstrates the capacity to interact with gamma-aminobutyric acid (GABA) receptors, potentially resulting in sedative and anti-anxiety effects. Chamomile also functions by stimulating the release of cortisol, has been found to alleviate anxiety. Previous studies have investigated the effects of this essential oil in various therapeutic contexts. A recent investigation carried out by (Ebrahimi et al., 2022) revealed the potential advantages associated with the use of chamomile essential oil aromatherapy in the reduction of anxiety levels among individuals having esophagogastroduodenoscopy. Additionally, this intervention was found to alleviate sensations of sorrow and improve the quality of sleep experienced by these patients. Currently, there is a lack of scholarly investigation about the concurrent utilization of lavender and chamomile essential oils by inhalation and its effects on reducing anxiety and pain in the field of pediatric dentistry.

Interestingly; The guidelines set forth by the American Academy of Pediatric Dentistry (AAPD) in 2023 suggest the utilization of aromatherapy as a non-pharmacological approach for alleviating anxiety and pain. Recommendations for Oral Health Policies The concept of endorsements refers to the act of publicly expressing support or approval for a person, According to Resources (The Reference Manual of Pediatric Dentistry 2022-2023 Definitions Oral Health Policies Recommendations Endorsements Resources, n.d.), the effectiveness and analgesic properties of lavender and chamomile oils have been the subject of previous research; yet, the majority of studies have mostly focused on adult populations. To the best of our current understanding, this research represents the inaugural investigation into the utilization of lavender oil inhalation as a means to examine the potential relationship between anxiety levels and vital signs in youngsters undergoing a stressful surgical dental intervention

ELIGIBILITY:
The inclusion criteria:

1. Patients with primary a mandibular molar that needs to be extracted.
2. Patients aged between 6 and 12 years.
3. Patients in their first dental visit.
4. Patients who are intellectually sufficient to complete the anxiety scale.
5. Children category 2, 3, 4 according to the Frankl Behaviour Rating Scale.
6. Patients whose parents were willing to participate in the study.

The exclusion criteria:

1. Patients with common allergies; Paediatric dental local anaesthesia allergies should be excluded to prevent bad reactions. Dental professionals should know how to treat local anaesthetic side effects such allergic and toxic responses. Consider the patient's medical history and physical condition before choosing a local anaesthetic dose and type. Identifying latex allergy patients and avoiding latex-containing products during dental operations is also important. For paediatric dental operations to be safe and effective, individuals with dental local anaesthesia allergies must be excluded.
2. Patients with respiratory tract infections or lung diseases; There is a potential increased susceptibility for paediatric patients to experience unfavourable respiratory tract effects following exposure to essential oils such as lavender and chamomile. The literature has demonstrated that upon inhalation, essential oils has the ability to effectively penetrate both the upper and lower regions of the respiratory tract
3. Patients with systemic problems; Lavender and chamomile essential oils may cause side effects in children with systemic diseases including impaired immune systems or chronic illnesses. Epidemiological studies have revealed no link between lavender essential oils and endocrine disturbance in youngsters. Children routinely exposed to these essential oils have similar endocrine abnormalities as those who are not .

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | immediately after the intervention
  Facial Image Scale (FIS) Score from (1-5) high score means worse outcome Score from (1-5) counting from left to right from 1 = not nervous at all to 5 = very very nervous
pain | immediately after the intervention
  Faces, legs ,activity ,cry , and consolability Score (0-10) high score means worse outcome

SECONDARY OUTCOMES:
Blood pressure (BP) | immediately after the intervention
  Sphygmomanometer
  mmHg
Pulse rate | immediately after the intervention
  Manual Beat/min
3. Oxygen saturation | immediately after the intervention
  Pulse oximeter Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Adel Albardisy, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebrahimi H, Mardani A, Basirinezhad MH, Hamidzadeh A, Eskandari F. The effects of Lavender and Chamomile essential oil inhalation aromatherapy on depression, anxiety and stress in older community-dwelling people: A randomized controlled trial. Explore (NY). 2022 May-Jun;18(3):272-278. doi: 10.1016/j.explore.2020.12.012. Epub 2021 Jan 9. PMID 33454232